CLINICAL TRIAL: NCT02059122
Title: Determination of Estimated Sensitivity for Dengue NS1 ELISAs
Brief Title: Sensitivity Study of Diagnostic for Early Detection of Dengue Infection
Status: Completed | Type: Observational
Sponsor: InBios International, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DSC0202/0093
Record Dates: First submitted 2014-02-07; First posted 2014-02-11 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Infectious Diseases
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — serum

SUMMARY:
This study is a multi-site trial assessing the sensitivity of DENV Detect™ NS1 ELISA versus standard reference tests (e.g. PCR or viral culture) for dengue diagnosis in the US and internationally.

The DENV Detect™ NS1 ELISA serves as an aid in the clinical laboratory diagnosis of early stages of Dengue infection in patients with clinical symptoms consistent with Dengue infection. This test is intended to be used on sera obtained within the first 7 days of symptoms. DENV Detect™ NS1 ELISA results (positive or negative) must be confirmed by testing with a reference standard test.

Subjects will be patients who present with symptoms consistent with dengue infection, such as fever and myalgia. After informed consent is obtained and the subject is screened for eligibility, 2 diagnostic samples will be collected. The first will be collected within the first 7 days of symptoms onset, and the second will be collected at least 7 days later, between the 10th and 21st days post-onset of symptoms.

ELISA and reference tests will be performed by different operators who are laboratory staff members. These staff members, blinded to each other's results, will evaluate the samples from each method independently.

ELIGIBILITY:
Inclusion Criteria:

* All age groups and both sexes.
* Initial serum samples must be collected within 1- 7 days of onset of symptoms consistent with Dengue virus infection.
* Information must be available about symptoms, age, and sex of patient from which samples are collected.
* The location of sample collection must be recorded.
* Archived samples that have been sent to reference labs for dengue or flavivirus testing should be considered for inclusion as test specimens in this study. If these specimens are included in this study, then they must have a documented history that the specimen was obtained within the first 7 days of onset of subject symptoms consistent with dengue infection.

Exclusion Criteria:

* Archived samples with linked personal identifiers or any sample for which personal information can be discovered.
* Prospective samples from nursing home residents; inmates/subjects in police custody; participants who are unable to understand verbal or written local language in which a certified translation of the informed consent is available, or requires a Legal Authorized Representative (LAR) for consent.
* Subject serum specimens that have undergone more than 2 freeze-thaw cycles or that have not been stored frozen.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Human males and females of varying ages and geographical locations where dengue fever is endemic. We will use retrospective (archived) and prospective human serum samples.
  Some study sites will only use retrospective (archived) serum samples not collected specifically for this study and not individually identifiable to the Investigators. These samples will fall under the category of "leftover" specimens as described by FDA guidance. These archived samples will have been collected from patients within 7 days after onset of symptoms consistent with Dengue infection.
  In addition paired prospective samples will be collected in compliance with human subject protection. The prospective samples will be collected from patients with symptoms consistent with Dengue infection. The first sample will be collected within the first 7 days of symptom onset; the second sample will be collected: 1) at least seven days later; and 2) between the 10th and 21st day of symptom onset.
Sampling Method: Probability Sample
Enrollment: 911 (Actual)
Dates: Start 2011-04; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
number of subjects with positive result | 1 day

CONTACTS AND LOCATIONS:
Locations (5):
- Universidad Nacional de Misiones (UNaM), Posadas, Argentina
- Leptospira Laboratory, Bridgetown, Barbados
- Universidad de Antioquia, Medellín, Colombia
- Ruhuna University, Galle, Sri Lanka
- AFRIMS, Bangkok, Thailand